CLINICAL TRIAL: NCT06005116
Title: Exploratory Study on the Effectiveness of Gallium [68Ga] NOTA-SGC8 Injection in the Staging of Bladder Cancer
Brief Title: [68Ga] NOTA-SGC8 in the Staging of Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIT-2022-0239
Record Dates: First submitted 2023-04-29; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; [68Ga]-NOTA-SGC8; PET/MR; Bladder Irrigation
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bladder Cancer Patients (Experimental)
  Interventions: Radiation: [68Ga]-NOTA-SGC8

INTERVENTIONS:
Radiation: [68Ga]-NOTA-SGC8 — Participants will be irrigated with [68Ga]-NOTA-SGC8 intravesically, with 0.05mCi/kg per person per time according to body weight, no more than 5mCi. The participants will be instructed to urinate cleanly before irrigation, and then irrigated [68Ga]-NOTA-SGC8 into the bladder via catheter for 30 minutes to make full contact between the injection and tumor. After 30 minutes, the injection will be withdrawn and 300ml normal saline will be injected into the bladder to maintain the shape of the bladder.

SUMMARY:
The goal of this clinical trial is to test the imaging and diagnostic ability of [68Ga]-NOTA-SGC8 PET/MR in bladder cancer patients with different stages. The main questions it aims to answer are:

* Tumor specific lighting ability of [68Ga]-NOTA-SGC8 in bladder cancer patients with different stages.
* The safety of [68Ga]-NOTA-SGC8. Participants will be irrigated with [68Ga]-NOTA-SGC8 into the bladder for tumor imaging under PET/MR. The imaging performance of [68Ga]-NOTA-SGC8 on different stages of bladder tumors will be systematically evaluated by combining with pathological sections of patients. Urine accumulation and radioactivity distribution of [68Ga]-NOTA-SGC8 will be measured. The adverse events will be recorded.

DETAILED DESCRIPTION:
Participants will be irrigated with [68Ga]-NOTA-SGC8 intravesically, with 0.05mCi/kg per person per time according to body weight, no more than 5mCi. The participants will be instructed to urinate cleanly before irrigation, and then irrigated [68Ga]-NOTA-SGC8 into the bladder via catheter for 30 minutes to make full contact between the injection and tumor. After 30 minutes, the injection will be withdrawn and 300ml normal saline will be injected into the bladder to maintain the shape of the bladder.

To evaluate the efficacy of [68Ga]-NOTA-SGC8 in imaging bladder tumors, the following indexes will be measured: specific imaging of the tumor area; specific imaging of its target PTK7 receptor protein; distribution in major organs; PET/MR imaging after administration; the absorbed dose of internal radiation based on the reference human hormone model using OLINDA software.

Tumor tissues of patients will be collected, and pathological sections of relevant patients will be analyzed after surgery. Immunohistochemistry will be used to verify the expression of PTK7 receptor in corresponding tumors. The association between PTK7 receptor protein and tumor malignancy, invasion, and stage will be evaluated by molecular imaging results.

All adverse events will be recorded within 24 hours after the administration of [68Ga]-NOTA-SGC8. Serious adverse events will be recorded for all subjects within 24 hours to 5 days after intravesical infusion. Blood and urine samples will be collected and the concentration of 68Ga-NOTA-SGC8 in the blood and urine will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed or previously diagnosed bladder tumors.
* At least one cystoscopy was performed within one month prior to enrollment, and the clinical diagnosis of bladder tumor was present.
* Age > 18 years, < 80 years
* Patients voluntarily participate and sign informed consent and are willing and able to follow protocol requirements.

Exclusion Criteria:

* Pregnancy, lactation, severe liver and kidney insufficiency and children;
* Participants who are allergic to the experimental drug, have an allergic disposition, or are allergic to multiple drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor specific lighting ability of [68Ga]-NOTA-SGC8 | 2 year
  Number of patients whose tumors are lightened under PET/MR with [68Ga]-NOTA-SGC8
Incidence of treatment-related adverse events of [68Ga]-NOTA-SGC8 | 2 year
  Adverse events within 24 hours of intravesical irrigation; Serious adverse events within 5 days of intravesical irrigation

SECONDARY OUTCOMES:
Staging ability of [68Ga]-NOTA-SGC8 | 2 year
  Accurate staging ability of [68Ga]-NOTA-SGC8 for bladder tumors
The expression of PTK7 in bladder tumor tissues | 2 year
  The expression of [68Ga]-NOTA-SGC8 target PTK7 receptor protein in bladder tumor tissues

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No